CLINICAL TRIAL: NCT07402486
Title: A Phase II Prospective Clinical Study to Evaluate the Feasibility, Safety, and Early Efficacy of Maastro Applicator High-Dose-Rate Brachytherapy in Selected Patients With Rectal Cancer
Brief Title: A Phase II Prospective Study of Maastro Applicator Brachytherapy for Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Wiwatchai Sittiwong, Dr., Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si1005/2568(IRB4)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
Keywords: HDR brachytherapy; Ractal cancer; Contact brachytherapy; MAASTRO applicator
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rectal HDR brachytherapy (Experimental): The patient will be given HDR brachytherapy via Maastro Applicator either as a monotherapy or boost
  Interventions: Radiation: Rectal HDR brachytherapy via Maastro Applicator

INTERVENTIONS:
Radiation: Rectal HDR brachytherapy via Maastro Applicator — Participants in this study will receive endorectal high-dose-rate (HDR) brachytherapy using the Maastro applicator as part of an organ-preserving treatment approach for rectal cancer.
  The Maastro applicator is a specially designed endorectal device intended for use with a standard HDR afterloading brachytherapy system (Ir-192 source). It enables delivery of a high, localized radiation dose directly to the rectal tumor with a steep dose fall-off, thereby minimizing radiation exposure to surrounding normal tissues.
  Procedure and delivery The brachytherapy procedure will be performed in a controlled procedural or operating room environment. Prior to treatment, patient identity, informed consent, and procedural safety checks will be confirmed. Local anesthesia and/or sedation will be administered according to institutional practice and patient needs.
  A rectoscope will be gently inserted to visualize the rectal lumen. Tumor localization and treatment geometry will be confirmed using direct

SUMMARY:
Rectal cancer is a common type of cancer and an important cause of illness and death worldwide. In 2020, cancers of the colon and rectum were the fourth most common cancers globally, and about one third of these cases were rectal cancer. Surgery is the main treatment for rectal cancer. In more advanced cases, chemotherapy and external beam radiotherapy are often given before surgery. However, surgery can sometimes result in a permanent stoma (an opening on the abdomen for bowel movements) and carries higher risks of complications, especially in older patients or those with other medical problems. Because of this, there is growing interest in treatment approaches that can control the cancer while avoiding major surgery when possible.

Some studies suggest that in carefully selected patients, rectal cancer can be treated without removing the rectum if the tumor responds well to radiation and chemotherapy. In these patients, survival outcomes may be similar to those who undergo surgery, although the risk of the cancer growing back locally can be slightly higher. This means that careful and long-term follow-up is very important. One of the key challenges with non-surgical treatment is determining how much radiation is needed to completely eliminate the tumor while minimizing side effects.

Contact X-ray brachytherapy is a type of radiation treatment that delivers a high dose of radiation directly to the tumor using low-energy X-rays. Because the radiation is given very close to the tumor, it can better target the cancer while reducing radiation exposure to surrounding healthy tissues. This technique has been used in Europe for many years and is recommended by international guidelines in selected patients, mainly within research settings. Other forms of brachytherapy using modern radiation sources can achieve similar dose distributions and may also support organ-preserving treatment strategies.

A new medical device called the Maastro applicator has been developed for use with high-dose-rate (HDR) brachytherapy systems. This applicator is designed to deliver radiation in a way that closely mimics low-energy X-ray treatments, while being compatible with widely available HDR brachytherapy equipment. Early technical studies suggest that it can deliver radiation accurately and safely, but its clinical effectiveness and safety in patients with rectal cancer have not yet been fully studied.

This phase II prospective study aims to evaluate the feasibility, safety, and early treatment outcomes of using the Maastro applicator for brachytherapy in patients with rectal cancer. The study will assess how often the tumor completely disappears after treatment, how well the cancer is controlled over time, the side effects of treatment, and how patients' quality of life changes. The results of this study will help determine whether this treatment approach is suitable for wider clinical use and will contribute to improving future treatment options for patients with rectal cancer.

DETAILED DESCRIPTION:
This is a single-center, Phase II prospective pilot study designed to evaluate the feasibility, safety, and early clinical outcomes of high-dose-rate (HDR) endorectal brachytherapy delivered using the Maastro applicator in patients with histologically confirmed rectal cancer.

Rectal cancer is commonly treated with surgery, frequently combined with chemotherapy and/or external beam radiotherapy (EBRT) in locally advanced disease. While surgery provides effective local control, it may be associated with substantial morbidity, including the risk of a permanent stoma and functional impairment. These concerns are particularly relevant in older patients or those with significant comorbidities. Consequently, there is increasing interest in organ-preserving strategies for selected patients who achieve a favorable response after non-operative treatment, provided that rigorous surveillance is maintained.

Contact-type local radiation boost approaches, including contact X-ray brachytherapy, deliver a high dose of radiation to the tumor with a steep dose gradient that limits dose to adjacent normal tissues. The Maastro applicator is a novel endorectal applicator developed for use with conventional HDR afterloading systems (Ir-192), intended to achieve a contact-like dose distribution using widely available HDR technology. Although dosimetric and simulation studies support its technical feasibility, prospective clinical evidence remains limited, motivating this Phase II evaluation.

Eligible participants will be adults (≥18 years) with rectal cancer whose tumors are accessible and suitable for endorectal HDR brachytherapy using the Maastro applicator, and who are deemed able to undergo the procedure with sedation/anesthesia as appropriate. Key exclusions include active inflammatory bowel disease (moderate-severe flare) or severe anorectal conditions that preclude safe applicator placement.

Participants will undergo standard baseline assessment per institutional practice, including clinical evaluation and appropriate imaging and/or endoscopic assessment. The Maastro applicator procedure will be performed in a controlled procedural environment. Tumor localization and applicator positioning will be guided by direct endoscopic visualization and transrectal ultrasound (TRUS) as applicable. HDR treatment plans (including applicator selection and relevant planning parameters) will undergo institutional verification and safety checks prior to delivery. Radiation will be delivered via an HDR afterloader through the applicator to the intended target volume. Patients will be observed post-procedure for immediate complications and provided standardized post-procedure instructions.

Participants will be followed at predefined intervals to assess tumor response, toxicity, and patient-reported outcomes. Tumor response will be assessed using clinical evaluation and imaging and/or endoscopy, with biopsy performed when clinically indicated. Adverse events will be captured and graded using CTCAE v5.0, including both acute and late gastrointestinal and genitourinary toxicities. Quality of life will be assessed longitudinally using validated instruments (EORTC QLQ-C30 and EORTC QLQ-CR29). Additional clinical endpoints include local control, regional control, progression-free survival, and overall survival. Exploratory analyses will assess associations between dosimetric parameters and tumor control and/or toxicity.

The primary endpoint is the clinical complete response rate following Maastro applicator HDR brachytherapy. Secondary endpoints include disease control outcomes (local/regional control, progression-free survival, overall survival), incidence of acute and late toxicities, and changes in quality of life over time. The planned sample size is 25 patients, consistent with a Phase II pilot cohort intended to generate early safety and efficacy signals and inform subsequent larger studies and protocol refinement.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years at the time of informed consent Histologically confirmed rectal cancer Any T, N, or M stage, provided the primary rectal lesion is suitable for endorectal HDR brachytherapy Tumor characteristics deemed suitable for treatment with the Maastro applicator (per investigator assessment) Rectal lesion accessible for applicator placement and adequate visualization Adequate organ function to undergo sedation/anesthesia and brachytherapy, as judged by the investigator Ability to comply with study procedures, imaging, and scheduled follow-up Written informed consent obtained prior to study participation

Exclusion Criteria:

Active inflammatory bowel disease with moderate to severe disease activity Uncontrolled proctitis not attributable to tumor involvement Severe anorectal conditions that preclude safe applicator placement (e.g., severe anal stenosis, uncontrolled hemorrhoidal bleeding, severe radiation-induced proctopathy in the target area) Any medical, psychiatric, or social condition that, in the opinion of the investigator, would interfere with safe study participation or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Complete Response (cCR) Rate | Within 6 months after completion of Maastro applicator HDR brachytherapy
  Clinical complete response is defined as the absence of detectable residual tumor within the treated rectal wall following Maastro applicator HDR brachytherapy, as determined by a combination of clinical examination, endoscopic assessment, and imaging (pelvic MRI), with biopsy performed when clinically indicated. Complete response requires no visible tumor, no ulceration suspicious for malignancy, and no radiologic evidence of residual disease at the treated site.

SECONDARY OUTCOMES:
Local Control Rate | Up to 2 years after completion of Maastro applicator HDR brachytherapy
  Local control is defined as the absence of tumor regrowth or persistence within the treated rectal wall or peri-rectal region (i.e., within the high-dose brachytherapy volume), as confirmed by clinical examination, endoscopy, and/or imaging (pelvic MRI), with biopsy performed when clinically indicated. Local failure is defined as biopsy-proven or radiologically evident local recurrence or progression at the treated site.
Regional Control Rate | Up to 2 years after completion of Maastro applicator HDR brachytherapy
  Regional control is defined as the absence of disease recurrence in regional lymphatic drainage areas of the rectum, including mesorectal, internal iliac, presacral, obturator, and external iliac lymph nodes, as assessed by imaging (MRI and/or PET/CT). Regional failure is defined as new or progressive nodal disease within these regions.
Progression-Free Survival (PFS) | Up to 2 years after initiation of Maastro applicator HDR brachytherapy
  Progression-free survival is defined as the time from the date of initiation of Maastro applicator HDR brachytherapy (or study enrollment) to the first documented evidence of disease progression (local, regional, or distant) or death from any cause, whichever occurs first. Patients alive without progression at last follow-up will be censored at that date.
Overall Survival (OS) | Up to 2 years after initiation of Maastro applicator HDR brachytherapy
  Overall survival is defined as the time from the date of initiation of Maastro applicator HDR brachytherapy (or study enrollment) to death from any cause. Patients alive at the time of analysis will be censored at the date of last follow-up.
Incidence of Acute and Late Treatment-Related Toxicities | From treatment initiation up to 2 years after completion of Maastro applicator HDR brachytherapy
  Treatment-related toxicities will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, including acute and late gastrointestinal and genitourinary toxicities. Acute toxicity is defined as events occurring within 90 days of treatment completion, and late toxicity as events occurring thereafter.
Quality of Life (QoL) | From baseline up to 2 years after completion of Maastro applicator HDR brachytherapy
  Quality of life will be evaluated using validated patient-reported outcome instruments, including the EORTC QLQ-C30 and EORTC QLQ-CR29 questionnaires. Changes from baseline will be analyzed over time.
Correlation of Dosimetric Parameters With Tumor Control and Toxicity | Up to 2 years after completion of Maastro applicator HDR brachytherapy
  Exploratory analyses will assess the association between dosimetric parameters of Maastro applicator HDR brachytherapy (e.g., prescribed dose, reference point dose, and treated volume) and clinical outcomes, including tumor control and treatment-related toxicities.

IPD SHARING:
Plan to Share IPD: Undecided